CLINICAL TRIAL: NCT04414956
Title: Clinical Usefulness of Combining Biomarkers (AFP, AFP-L3, and PIVKA-II) With Abdominal Sonography or Computed Tomography for Early Detection of Hepatocellular Carcinoma
Brief Title: Combining Biomarkers (AFP, AFP-L3, and PIVKA-II) and Image Tools for Early Detection of Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: Korea University Ansan Hospital (Other); Soonchunhyang University Hospital (Other); Korea University Guro Hospital (Other); The Catholic University of Korea (Other); Samsung Medical Center (Other); Asan Medical Center (Other); Korea University Anam Hospital (Other); Keimyung University Dongsan Medical Center (Other); Severance Hospital (Other); Hanyang University (Other); Konkuk University Hospital (Other); Seoul National University Hospital (Other); Inje University (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Soon Ho Um, Professor, Korea University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HCCAFPL3
Record Dates: First submitted 2020-05-20; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma; Surveillance
Keywords: Liver Cirrhosis; Hepatocellular Carcinoma; Surveillance; AFP-L3; AFP; PIVKA-II; Sonography; CT
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular | interventions — Ultrasonography; Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: Patients with cirrhosis will receive the surveillance test using three biomarker tests and sonography every six months and contrast-enhanced CT annually
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surveillance (Other): All participants will be examined with three biomarker tests and sonography every six months and contrast-enhanced CT annually.
  Interventions: Diagnostic Test: AFP-L3; Diagnostic Test: AFP; Diagnostic Test: PIVKA-II; Diagnostic Test: Sonography; Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: AFP-L3 — AFP-L3 will be tested using serum sample every 6 months.
  Other Names: Lens culinaris agglutinin-reactive fraction of AFP
Diagnostic Test: AFP — AFP will be tested using serum sample every 6 months.
  Other Names: Alpha fetoprotein
Diagnostic Test: PIVKA-II — PIVKA-II will be tested using serum sample every 6 months.
  Other Names: Protein induced by vitamin K absence or antagonist-II; des-gamma-carboxy prothrombin
Diagnostic Test: Sonography — Sonography will be tested by experts every 6 months.
  Other Names: Ultrasound; US
Diagnostic Test: CT — Contrast-enhanced CT will be tested annually.
  Other Names: Computed tomography

SUMMARY:
In this study, three biomarkers tests (AFP, AFP-L3 and PIVKA-II) and abdominal sonography or CT scans are performed every 6 months to detect hepatocellular carcinoma (HCC) early in patients with cirrhosis, a high-risk group of HCC. The aim of this study is to confirm the early HCC diagnosis rate in patients with cirrhosis and compare the detection efficacy between tests.

DETAILED DESCRIPTION:
Early diagnosis of HCC is the most important factor in improving the prognosis of the disease. A surveillance test for early diagnosis of HCC in Korea is to perform alfa fetoprotein (AFP) and abdominal sonography every 6-months in high-risk groups. However, the detection rate of HCC using AFP and abdominal sonography is very low. There are several reports that the combination of the multiple biomarker tests including AFP, AFP L3, and PIVKA-II increased the early HCC detection only one test. Therefore, in the surveillance test for HCC, the combination of three tests with sonography would be helpful in the early diagnosis of HCC. However, there was few prospective large-scale studies about this issue.

Compared with abdominal sonography, contrast-enhanced CT or MRI is more useful in finding intrahepatic lesions of liver cirrhosis. However, there is no evidence data on combining sono/CT and biomarkers could improve the diagnosis for early HCC. Thus, it is essential to verify this prospectively in the real clinical practices to make recommendations based on a high level of evidence in the future. The investigators are conducting a prospective study which examines three biomarker tests and sonography every six months and contrast-enhanced CT annually for HCC surveillance in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis meeting one of the followings:

  i. Histologically confirmed liver cirrhosis ii. Imaging findings with liver cirrhosis (liver surface undulation, irregularity, or nodularity by US, CT, or MRI) plus one of followings: liver stiffness measurement ≥ 12.5 kilopascal, esophago-gastric varices, thrombocytopenia (<120,000/mm3), hypoalbuminemia (<3.5 g/dL), splenomegaly ≥12 cm) iii. Imaging findings with liver cirrhosis together with biomarkers suggesting liver cirrhosis (APRI ≥2.0 or fibrosis-4 ≥3.6) iv. Imaging findings with liver cirrhosis with history of hepatic decompensation (ascites, esophago-gastric variceal bleeding, jaundice, hepatic encephalopathy))
* Expected survival more than 1 year
* Child Pugh score 5-10 at the time of enrollment
* Serum creatinine ≤1.5mg/dL
* Age between 19 and 75 years old
* No significant underlying medical illness affecting patient's survival
* Patients available for regular follow-up according to the study protocol

Exclusion Criteria:

* History of HCC
* AFP >20 ng/mL
* Hepatic nodule ≥ 1 cm by US or CT Exceptionally, nodules showing characteristic features of benign lesion such as hemangioma or pathologically conformed benign lesion are permitted for study inclusion.
* Hepatic nodule less than 1 cm on US but imaging findings suggesting HCC by contrast enhanced US, CT, or MRI
* Child-Pugh score ≥ 11
* History of liver transplantation
* Expecting liver transplantation within 1 year
* Hypersensitivity on CT contrast dye
* Any contraindication for CT
* Not able to perform abdominal US
* Other uncontrolled malignancy
* Patients taking warfarin

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1418 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
HCC occurrence | 3 years after enrollment
  Detection of HCC occurrence by three biomarkers and two image modalities

SECONDARY OUTCOMES:
Early HCC occurrence | 3 years after enrollment
  Detection of HCC less than 2cm

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - The Catholic University of Korea Uijeongbu St.Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Inje University SangGye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St.Mary's Hospital, Seoul
  - Chung-Ang University Hosptial, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Serag HB. Hepatocellular carcinoma. N Engl J Med. 2011 Sep 22;365(12):1118-27. doi: 10.1056/NEJMra1001683. No abstract available. PMID 21992124
- [Background] Korean Liver Cancer Study Group (KLCSG); National Cancer Center, Korea (NCC). 2014 KLCSG-NCC Korea Practice Guideline for the Management of Hepatocellular Carcinoma. Gut Liver. 2015 May 23;9(3):267-317. doi: 10.5009/gnl14460. PMID 25918260
- [Background] Yim HJ, Suh SJ, Um SH. Current management of hepatocellular carcinoma: an Eastern perspective. World J Gastroenterol. 2015 Apr 7;21(13):3826-42. doi: 10.3748/wjg.v21.i13.3826. PMID 25852267
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Result] Yim SY, Seo YS, Jung CH, Kim TH, Lee JM, Kim ES, Keum B, Jong YK, An H, Kim JH, Yim HJ, Kim DS, Jeen YT, Yeon JE, Lee HS, Chun HJ, Byun KS, Um SH, Kim CD, Ryu HS. The management and prognosis of patients with hepatocellular carcinoma: what has changed in 20 years? Liver Int. 2016 Mar;36(3):445-53. doi: 10.1111/liv.12960. Epub 2015 Oct 12. PMID 26352789
- [Result] Sterling RK, Jeffers L, Gordon F, Venook AP, Reddy KR, Satomura S, Kanke F, Schwartz ME, Sherman M. Utility of Lens culinaris agglutinin-reactive fraction of alpha-fetoprotein and des-gamma-carboxy prothrombin, alone or in combination, as biomarkers for hepatocellular carcinoma. Clin Gastroenterol Hepatol. 2009 Jan;7(1):104-13. doi: 10.1016/j.cgh.2008.08.041. Epub 2008 Sep 17. PMID 18849011
- [Result] Taketa K, Sekiya C, Namiki M, Akamatsu K, Ohta Y, Endo Y, Kosaka K. Lectin-reactive profiles of alpha-fetoprotein characterizing hepatocellular carcinoma and related conditions. Gastroenterology. 1990 Aug;99(2):508-18. doi: 10.1016/0016-5085(90)91034-4. PMID 1694805
- [Result] Taketa K, Endo Y, Sekiya C, Tanikawa K, Koji T, Taga H, Satomura S, Matsuura S, Kawai T, Hirai H. A collaborative study for the evaluation of lectin-reactive alpha-fetoproteins in early detection of hepatocellular carcinoma. Cancer Res. 1993 Nov 15;53(22):5419-23. PMID 7693340
- [Result] Oka H, Saito A, Ito K, Kumada T, Satomura S, Kasugai H, Osaki Y, Seki T, Kudo M, Tanaka M; Collaborative Hepato-Oncology Study Group of Japan. Multicenter prospective analysis of newly diagnosed hepatocellular carcinoma with respect to the percentage of Lens culinaris agglutinin-reactive alpha-fetoprotein. J Gastroenterol Hepatol. 2001 Dec;16(12):1378-83. doi: 10.1046/j.1440-1746.2001.02643.x. PMID 11851836
- [Result] Nakamura S, Nouso K, Sakaguchi K, Ito YM, Ohashi Y, Kobayashi Y, Toshikuni N, Tanaka H, Miyake Y, Matsumoto E, Shiratori Y. Sensitivity and specificity of des-gamma-carboxy prothrombin for diagnosis of patients with hepatocellular carcinomas varies according to tumor size. Am J Gastroenterol. 2006 Sep;101(9):2038-43. doi: 10.1111/j.1572-0241.2006.00681.x. Epub 2006 Jul 18. PMID 16848811
- [Result] Choi JY, Jung SW, Kim HY, Kim M, Kim Y, Kim DG, Oh EJ. Diagnostic value of AFP-L3 and PIVKA-II in hepatocellular carcinoma according to total-AFP. World J Gastroenterol. 2013 Jan 21;19(3):339-46. doi: 10.3748/wjg.v19.i3.339. PMID 23372355
- [Result] Yoon YJ, Han KH, Kim DY. Role of serum prothrombin induced by vitamin K absence or antagonist-II in the early detection of hepatocellular carcinoma in patients with chronic hepatitis B virus infection. Scand J Gastroenterol. 2009;44(7):861-6. doi: 10.1080/00365520902903034. PMID 19391065
- [Result] Seo SI, Kim HS, Kim WJ, Shin WG, Kim DJ, Kim KH, Jang MK, Lee JH, Kim JS, Kim HY, Kim DJ, Lee MS, Park CK. Diagnostic value of PIVKA-II and alpha-fetoprotein in hepatitis B virus-associated hepatocellular carcinoma. World J Gastroenterol. 2015 Apr 7;21(13):3928-35. doi: 10.3748/wjg.v21.i13.3928. PMID 25852278
- [Result] Lim TS, Kim DY, Han KH, Kim HS, Shin SH, Jung KS, Kim BK, Kim SU, Park JY, Ahn SH. Combined use of AFP, PIVKA-II, and AFP-L3 as tumor markers enhances diagnostic accuracy for hepatocellular carcinoma in cirrhotic patients. Scand J Gastroenterol. 2016 Mar;51(3):344-53. doi: 10.3109/00365521.2015.1082190. Epub 2015 Sep 4. PMID 26340708
- [Result] Di Martino M, De Filippis G, De Santis A, Geiger D, Del Monte M, Lombardo CV, Rossi M, Corradini SG, Mennini G, Catalano C. Hepatocellular carcinoma in cirrhotic patients: prospective comparison of US, CT and MR imaging. Eur Radiol. 2013 Apr;23(4):887-96. doi: 10.1007/s00330-012-2691-z. Epub 2012 Nov 18. PMID 23179521
- [Result] Kudo M, Matsui O, Izumi N, Iijima H, Kadoya M, Imai Y, Okusaka T, Miyayama S, Tsuchiya K, Ueshima K, Hiraoka A, Ikeda M, Ogasawara S, Yamashita T, Minami T, Yamakado K; Liver Cancer Study Group of Japan. JSH Consensus-Based Clinical Practice Guidelines for the Management of Hepatocellular Carcinoma: 2014 Update by the Liver Cancer Study Group of Japan. Liver Cancer. 2014 Oct;3(3-4):458-68. doi: 10.1159/000343875. PMID 26280007
- [Result] Chou R, Cuevas C, Fu R, Devine B, Wasson N, Ginsburg A, Zakher B, Pappas M, Graham E, Sullivan SD. Imaging Techniques for the Diagnosis of Hepatocellular Carcinoma: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 May 19;162(10):697-711. doi: 10.7326/M14-2509. PMID 25984845